CLINICAL TRIAL: NCT04816006
Title: Enhancing Cognitive Function in Breast Cancer Survivors Through Community-based Exercise Training
Brief Title: Breast Cancer, Reasoning, and Activity Intervention
Acronym: BRAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Diane K. Ehlers, Ph.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MC231001; 23-000020 (Other: Mayo Clinic Institutional Review Board); 852-20-FB (Other: Previous IRB); R37CA252060 (NIH); NCI-2021-09939 (Registry Identifier: Clinical Trials Reporting Program)
Record Dates: First submitted 2021-02-26; First posted 2021-03-25 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Breast Neoplasms; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Cancer-related Cognitive Dysfunction
Keywords: physical activity; exercise; cognition; brain health; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Aerobic Exercise) (Experimental): Patients attend 3 weekly exercise sessions over 60-75 minutes per week in weeks 1-2, 2 sessions over 70-70 each week in weeks 3-4, 1 session over 90-120 minutes each week in weeks 5-8, biweekly sessions over 120-150 per week across weeks 9-16, and monthly sessions over at least 150 minutes per week in weeks 17-24 for a total of 20 supervised sessions. Patients undergo MRI and wear an accelerometer throughout the study.
  Interventions: Behavioral: Aerobic Exercise Training
- Arm II (Health Education) (Active Comparator): Patients participate in up to 9 monthly classes/webinars. Patients also receive informational pdfs, videos, and/or podcasts, and a one-year subscription to the Mayo Clinic Health Letter. Patients undergo a gait assessment and MRI, as well as wear an accelerometer throughout the study.
  Interventions: Other: Health Education (Active comparator)

INTERVENTIONS:
Behavioral: Aerobic Exercise Training — Breast cancer survivors in the intervention group will participate in a 24-week moderate intensity exercise program led by community-based fitness center personal trainers. Individually-tailored exercise prescriptions will be developed based upon each participant's baseline maximal graded exercise test (heart rate corresponding with %VO2 peak) and symptom limitation. Sessions will be progressive in nature such that the volume of exercise increases across weeks. Treadmill walking is the primary mode of exercise. However, participants will be permitted to use other cardiovascular equipment (e.g., elliptical machines, stationary bicycles) as prescribed by their exercise trainer. The trainer will supervise three weekly exercise sessions in Weeks 1-2, two in Weeks 3-4, one in Weeks 5-8, biweekly across weeks 9-16, and monthly in Weeks 17-24 (N=20 supervised sessions).
  Arms: Arm I (Aerobic Exercise)
Other: Health Education (Active comparator) — Breast cancer survivors in the Health Education group will participate in education sessions with a health educator and receive monthly newsletters/webinars (N=20 total contacts) across 24 weeks. The program will include cancer support and discussion of cancer-related wellness topics (e.g., stress management, coping). Control group participants will be offered a 6-month fitness center membership upon study completion.
  Other Names: Control Group
  Arms: Arm II (Health Education)

SUMMARY:
This phase II trial tests whether an exercise intervention works to improve cognitive function in breast cancer survivors. Many breast cancer survivors report cancer-related cognitive impairment, which this has recently become a priority in clinical research due to its dramatic impact on daily functioning, quality of life, and long-term health. Aerobic exercise has the potential to improve cognitive function and brain health in older adults and is recommended as a safe, tolerable, and accessible complementary therapy for breast cancer survivors. This study aims to understand the effects of physical activity compared with health education on memory, attention, and brain health in women with breast cancer. Study findings may help researchers design more programs that can improve memory, attention, and brain health in other women with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the effectiveness of a 6-month, community-based aerobic exercise intervention on multiple indicators of cognitive function in breast cancer survivors (BCS) aged 50 and older (N=160).

II. Gather information on the intervention's potential for scalability using the Reach Effectiveness Adoption Implementation Maintenance (RE-AIM) framework.

EXPLORATORY OBJECTIVES:

I. Explore potential moderators and mediators of the effects of aerobic exercise training on cognitive function.

II. Investigate the feasibility of urinary metabolites as biomarkers of overall diet patterns.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients attend 3 weekly exercise sessions over 60-75 minutes per week in weeks 1-2, 2 sessions over 70-70 each week in weeks 3-4, 1 session over 90-120 minutes each week in weeks 5-8, biweekly sessions over 120-150 per week across weeks 9-16, and monthly sessions over at least 150 minutes per week in weeks 17-24 for a total of 20 supervised sessions. Patients undergo a gait assessment and magnetic resonance imaging (MRI), as well as wear an accelerometer throughout the study.

ARM II: Patients participate in up to 9 monthly classes/webinars. Patients also receive informational portable document format (pdfs), videos, and/or podcasts, and a one-year subscription to the Mayo Clinic Health Letter. Patients undergo a gait assessment and MRI, as well as wear an accelerometer throughout the study.

After completion of study intervention, patients are followed up with at 6 months.

ELIGIBILITY:
Inclusion Criteria

* PRE-REGISTRATION: Age ≥50 years at time of pre-registration visit according to participant report and/or clinical determination
* PRE-REGISTRATION: First, primary diagnosis of stage I-IIIa breast cancer according to participant report and/or clinical determination
* PRE-REGISTRATION: Post-surgery and completed primary treatment (i.e., surgery, chemotherapy, and/or radiation therapy) 3-36 months prior to registration according to participant report and/or clinical determination
* PRE-REGISTRATION: Sedentary except for casual lifestyle recreation defined as self-reporting no more than 90 minutes per week of moderate-intensity aerobic exercise within the last 6 months
* PRE-REGISTRATION: Self-reported ability to complete assessments by themselves or with assistance
* REGISTRATION: Age ≥50 years as confirmed via clinical determination
* REGISTRATION: Able to provide medical record release to confirm eligibility
* REGISTRATION: First, primary diagnosis of stage I-IIIa breast cancer as confirmed via clinical determination
* REGISTRATION: Post-surgery and completed primary treatment (i.e., surgery, chemotherapy, and/or radiation therapy) 3-36 months prior to pre-registration as confirmed via clinical determination
* REGISTRATION: No evidence of possible cognitive impairment as assessed using the Telephone Interview of Cognitive status (13-item modified version) (TICS-M; score > 21) NOTE: Only individuals who pass the TICS-M during pre-registration will be invited to participate in the urine substudy
* REGISTRATION: Receive physician's clearance to participate in an exercise program

NOTE: Individuals with conditions/diagnoses deemed important by the primary investigator will be required to provide clearance for exercise from their cardiologist. Example conditions include:

* History of major multiple myocardial infarctions (MI)
* Recent electrocardiogram (ECG) changes or recent MI
* Resting or unstable angina
* Significant multivessel coronary occlusion (≥ 70%) on angiography
* Uncontrolled and/or serious arrhythmias
* 3rd degree heart block
* Acute congestive heart failure or ejection fraction < 30%

  * REGISTRATION: Ability to complete assessments by themselves or with assistance

Exclusion Criteria:

* PRE-REGISTRATION: Stage 0 breast cancer diagnosis OR metastatic disease
* PRE-REGISTRATION: Currently receiving or < 3 months since receiving chemotherapy or radiation therapy for cancer, or greater than 36 months post primary treatment
* PRE-REGISTRATION: Planned surgery during the intervention period
* PRE-REGISTRATION: Second cancer diagnosis (excluding non-invasive skin cancers or carcinoma-in-situ for any cancer)
* PRE-REGISTRATION: Unable to travel regularly to the study locations for intervention sessions and data collection
* PRE-REGISTRATION: Unwilling to return to enrolling institution for follow-up
* PRE-REGISTRATION: Self-reported inability to walk without assistance or devices
* REGISTRATION: History of stroke, transient ischemic attack, other neurological disorders, or brain surgery involving tissue removal as confirmed via clinical determination
* REGISTRATION: Clinically significant TICS-M score (< 21) during baseline procedures
* REGISTRATION: Not able to provide physician re-clearance for exercise if required based upon clinically significant baseline exercise test (as determined by ECG and blood pressure monitoring)
* REGISTRATION: Contraindications to functional magnetic resonance imaging (fMRI) in accordance with the Mayo Clinic Department of Radiology safety protocols
* REGISTRATION: Clinically significant MRI scan as determined by physician review in which the following is advised via radiologist overread: remarkable/abnormal limited diagnostic brain image with recommended medical follow-up
* REGISTRATION: Enrolled in another physical activity program
* REGISTRATION: Unable to walk without assistance or devices
* REGISTRATION: Unwilling to complete study requirements
* REGISTRATION: Unwilling to be randomized to the exercise group or health education group
* REGISTRATION: Unable or unwilling to continuously wear and regularly sync/charge an activity tracker during the study period
* REGISTRATION: Unable to travel regularly to the study locations for intervention sessions and data collection
* REGISTRATION: Unwilling to return to enrolling institution for follow-up

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in inhibitory control | baseline (Month 0), post-intervention (month 6), follow up (month 12)
  Change in interference score on Stroop task, with positive values indicating greater inhibitory control.
Change in cognitive flexibility | baseline (Month 0), post-intervention (month 6), follow up (month 12)
  Change in accuracy on Shifting Attention task, with higher values indicating greater cognitive flexibility
Change in executive function processing | baseline (Month 0), post-intervention (month 6), follow up (month 12)
  Change in reaction time on Shifting Attention task, with lower values indicating greater cognitive flexibility
Change in short-term memory | baseline (Month 0), post-intervention (month 6), follow up (month 12)
  Change in accuracy on Visual Memory task, with higher accuracy indicating greater short-term memory
Change in verbal memory | baseline (Month 0), post-intervention (month 6), follow up (month 12)
  Change in number recalled on Hopkins Verbal Learning task, with higher values indicating greater verbal memory
Change in working memory | baseline (Month 0), post-intervention (month 6), follow up (month 12)
  Change in reaction time the 4-part Continuous Performance task, with lower values indicating greater working memory
Change in brain volume | baseline (Month 0), post-intervention (month 6)
  Change in mean cortical thickness of brain regions of interest as measured by an anatomic MRI brain scan
Change in white matter integrity | baseline (Month 0), post-intervention (month 6)
  Change in fractional anisotropy as measured by diffusion MRI.
Change in resting state functional connectivity | baseline (Month 0), post-intervention (month 6)
  Change in within-network pairwise correlation estimates as measured using a multiband echo planar imaging (mb-EPI) functional MRI sequence
Change in self-reported cognitive function | baseline (Month 0), post-intervention (month 6), follow up (month 12)
  The perceived cognitive impairments subscale of the Functional Assessment in Cancer Therapy - Cognition (FACT-Cog) will be used to measure self-reported cognition. Scores range from 0-72, with higher scores indicating better cognitive function.
Reach | baseline (Month 0)
  Participation rate among eligible individuals contacted about the study.
Adoption | post-intervention (month 6)
  Sociodemographics questionnaire to describe demographics characteristics and experience among personal trainers
Change in Cardiorespiratory Fitness | baseline (Month 0), post-intervention (month 6), follow up (month 12)
  Change in Peak VO2 as measured by a modified Balke treadmill graded exercise test protocol.
Change in Cancer-related Fatigue | baseline (Month 0), post-intervention (month 6), follow up (month 12)
  The Functional Assessment in Chronic Illness Therapy (FACIT) - Fatigue Scale will be used to measure cancer-related fatigue. Scores range from 0-52, with higher scores indicating less cancer-related fatigue.
Implementation | post-intervention (month 6)
  Percent of session checklist items completed as intended
Maintenance | follow up (month 12)
  The number of participants who withdraw during the follow-up period.
Change in processing speed | baseline (Month 0), post-intervention (month 6), follow up (month 12)
  Change in reaction time on Symbol Digit Coding task, with lower values indicating greater processing speed
Change in attention | baseline (Month 0), post-intervention (month 6), follow up (month 12)
  Change in choice reaction time on Continuous Performance task, with lower values indicating greater sustained attention

CONTACTS AND LOCATIONS:
Overall Officials: Diane K. Ehlers, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Although the final dataset will not include identifying information, there is still a possibility of deductive disclosure of identity. Therefore, data will not be shared via an NIH or approved public repository; however, we will share de-identified data as required for publication in scientific journals and with outside collaborators and scientists upon request.
Supporting Information: Study Protocol
Time Frame: Data will be shared via scientific journals at the time of publication and with outside collaborators before publication.
Access Criteria: We will make data available to researchers who agree to use the data only for research purposes, protect the data using secure computer technologies, and destroy the data after relevant analyses are completed and manuscripts published.

REFERENCES:
- [Derived] Ehlers DK, Austin JD, Ernst B, Page LL, Ofori E, Porter GC, Fanning J, Hickman G, McKim P, Cole M, Donaldson M, Braden BB, Kunze KL, Butterfield RJ, Baxter LC, Ahles TA, Estabrooks P. Enhancing cognitive function in breast cancer survivors through community-based aerobic exercise training: protocol for a Hybrid Type I effectiveness-implementation study employing a randomised controlled design. BMJ Open. 2025 Jul 13;15(7):e104378. doi: 10.1136/bmjopen-2025-104378. PMID 40659404
- See also: Mayo Clinic Clinical Trials: Breast Cancer, Reasoning, and Activity Intervention — https://www.mayo.edu/research/clinical-trials/cls-20558432